CLINICAL TRIAL: NCT05816486
Title: Longitudinal Observational Study to Determine the Correlation Between Patient's Pharmacodynamic Response to Immunosuppressants Measured in Vitro With IMMUNOBIOGRAM and of Rejection in Graft Biopsies in Patients With Renal Transplantation
Brief Title: BIOtechnology Applied to Renal TRansplantation With IMmunobiogram
Acronym: BIOTRAIM
Status: Completed | Type: Observational
Sponsor: Biohope Scientific Solutions for Human Health, S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: BH-IMBG-TR-2021
Record Dates: First submitted 2023-02-09; First posted 2023-04-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Kidney Transplant Failure and Rejection
Keywords: Kidney Transplant Rejection; Immunosuppression; Immune cell bioassay; Pharmacodynamics; Oportunistic infections
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Renal biopsy and blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Prospective - Longitudinal: Longitudinal follow-up cohort in which all patients who are going to receive a kidney transplant and meet the selection criteria for this study cohort will be included. This cohort will be recruited at sites that routinely perform Protocol Biopsies (PB) one year after transplant. A pre-transplant and post-transplant follow-up IMBG at 3, 6, 9 and 12 months will be performed, and additional IMBG will be carried out when an indication biopsy is required due to a suspected rejection during the patients' follow-up. A protocol biopsy will be performed after one year of follow-up of the patients.
  Interventions: Diagnostic Test: Immunobiogram
- Cross-sectional: Patients in whom an Indication Biopsy (IB) is to be performed due to suspicion of rejection. This cohort may be recruited in all sites participating in the study, including sites where annual protocol biopsies are not routinely performed. An IMBG will be performed coinciding with the IB. This cohort will include patients who have had their transplant for less than 5 years.
  Interventions: Diagnostic Test: Immunobiogram
- Control: Patients who have received a kidney transplant or a re-transplant less than 5 years before inclusion in the study and have shown a stable clinical course after 6 months from the RT, defined as: patients without previous rejection episodes nor indication biopsies, who do not show signs of renal impairment and are dnDSA negative, without changes in immunosuppressive drugs in the last 6 weeks and without opportunistic infections in the last six months before entering in the study. An IMBG will be performed coinciding with the only visit.
  Interventions: Diagnostic Test: Immunobiogram

INTERVENTIONS:
Diagnostic Test: Immunobiogram — This is not an interventional study. However the assay being tested on the blood samples of all enrolled participants is the Immunobiogram (IMBG). IMBG is an in vitro diagnostic immunoassay which can obtain dose-response curves that describe the inhibitory effect of each immunosuppressant on immune response cells (immunologically stimulated PBMCs) in kidney transplant patients.

SUMMARY:
Immunobiogram (IMBG) is a novel in vitro diagnostic bioassay developed by Biohope Scientific Solutions for Human Health SL, that allows to measure the pharmacodynamic response to individual immunosuppressive drugs in patients with a renal transplantation. Pharmacodynamics can complement the already available pharmacokinetic information on immunosuppressants and enable a more individualized evaluation of the immunosuppressive therapy.

The aim of this study is to evaluate the association between the pharmacodynamic response to individual immunosuppressants taken by the patient measured in vitro with IMBG and the existence of signs of graft rejection in biopsies (upon indication or protocol) performed in a sample of kidney transplant patients.

The main hypothesis is that a lower sensitivity to the immunosuppressive drugs taken by the patient will be associated with a higher probability of rejection.

DETAILED DESCRIPTION:
Immunobiogram (IMBG) is a novel bioassay that allows to measure in vitro the inhibitory effect of a battery of individual immunosuppressants on the patient's immune cells (immunologically stimulated PBMCs).

Studies conducted in kidney transplant patients have shown that IMBG is a valid and accurate instrument, capable of determining each patient's pharmacodynamic response profile to individual immunosuppressive drugs.

Health professionals who monitor kidney transplant patients currently have information only on immunosuppressant pharmacokinetics to adjust the regimen of the immunosuppressants they use to treat the patients to avoid graft rejection. The pharmacodynamic measurement of the in vitro effect of each immunosuppressant in the patient could complement the pharmacokinetic information and enable more personalized approaches.

The main objective of this study is to evaluate the association between the pharmacodynamic response to individual immunosuppressants taken by the patient measured with IMBG and the existence of signs of graft rejection in biopsies (upon indication or protocol) performed in a sample of kidney transplant patients.

A longitudinal follow-up cohort of patients will be recruited from prior to the transplant (at sites that regularly perform a protocol graft biopsy after a year) and a cross-sectional cohort of patients will also be included when an indication biopsy is performed during the first five years after kidney transplantation due to a suspicion of rejection at sites that do not routinely perform protocol biopsies.

Given that one of the main challenges that clinicians face in the follow-up of patients is to reduce the risk of renal graft rejection, while minimizing the incidence of secondary effects related to immunosuppressive therapy, it is proposed as a secondary objective to evaluate in the longitudinal cohort the incidence of "therapeutical failure" due to graft failure or due to the appearance of serious adverse effects attributable to immunosuppression and analyze its relationship with the profile of sensitivity to immunosuppressants taken by the patient measured with IMBG.

It will be also evaluated if the IMBG sensitivity to immunosuppressive drugs measured pretransplant predict the ocurrence of rejection or adverse events during the first year postransplant.

Finally, the changes over time presented by the IMBG in various determinations and the correlation between IMBG results and other lymphocyte activation parameters obtained by flow cytometry will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

Longitudinal cohort:

1. Patients > 18 years of age.
2. Candidate to receive a kidney transplant or re-transplant.
3. Patients in whom it is planned to routinely perform a protocol biopsy one year after the kidney transplant for which there is no contraindication at the time of inclusion in the study.
4. Patients in whom a pre-transplant blood sample can be drawn that is viable for the processing of an IMBG.
5. Patients who give their written informed consent to participate in the study.

Cross-sectional cohort:

1. Patients > 18 years of age.
2. Patients who have received a kidney transplant or re-transplant less than 3 years before inclusion in the study.
3. Patients in whom an indication biopsy is to be performed due to suspicion of rejection.
4. Patients in whom a blood sample can be drawn in a period of time less than 8 days before or after the Indication Biopsy that is viable for the processing of an IMBG.
5. Patients who give their written informed consent to participate in the study.

Exclusion Criteria (PROSPECTIVE AND CROSS-SECTIONAL COHORT):

1. Patient with a double transplant (kidney + other organ).
2. Contraindication for performing a renal graft biopsy.
3. Active autoimmune diseases in the 12 months prior to the study visit (with systemic inflammatory exacerbation in the year prior to study inclusion, despite immunosuppressive therapy).
4. Very elderly cadaver donor transplant (>80 years of age).
5. Donors in asystole II.
6. Recurrent primary kidney disease in the case of primary focal and segmental hyalinosis or hemolytic-uremic syndrome.
7. Active HIV, HBV or HCV infection or other severe infections (to prevent risks in the processing of samples in conventional laboratories).
8. Concomitant medical conditions that may affect the patient's participation in the study.

Control cohort:

Inclusion criteria:

1. Patients > 18 years of age.
2. Patients who have received a kidney transplant or re-transplant less than 5 years before inclusion in the study.
3. A stable course after 6 months post-transplant defined as:

   * Lack of renal impairment (GFR > 50 ml/min/1.73 m2 and proteinuria < 300 mg/g)
   * No previous rejection episodes and no graft indication biopsies
   * No positive dnDSA
   * No change in the active principle of immunosuppressive drugs in the last 6 weeks
   * No opportunistic infections in the last 6 months
4. Patients in whom a blood sample can be drawn suitable for IMBG processing.
5. Patients (or their legal representative) who give their written informed consent to participate in the study.

Exclusion criteria:

1. Patient with a double transplant (kidney + other organ).
2. Active autoimmune diseases in the 12 months prior to the study visit (with systemic inflammatory exacerbation in the year prior to study inclusion, despite immunosuppressive therapy).
3. Very elderly cadaver donor transplant (>80 years of age).
4. Donors in asystole II.
5. Recurrent primary kidney disease in the case of primary focal and segmental hyalinosis or hemolytic-uremic syndrome.
6. Active HIV, HBV or HCV infection or other severe infections (to prevent risks in the processing of samples in conventional laboratories).
7. Concomitant medical conditions that may affect the patient's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Prospective longitudinal cohort: all patients who are to receive a kidney transplant and meet the screening criteria for this study cohort. This cohort will be recruited in sites that routinely perform a Protocol Biopsy (PB) one year after transplant.
  2. Cross-sectional cohort: patients in whom an Indication Biopsy (IB) is to be performed due to suspicion of rejection. This cohort may be recruited in all sites participating in the study and patients will be enrolled competitively.
  3. Control cohort: cross-sectional cohort to include patients who have received a kidney transplant or a re-transplant less than 5 years before inclusion in the study and have shown a stable clinical course after 6 months post-transplant. An IMBG will be performed coinciding with the study visit.
Sampling Method: Probability Sample
Enrollment: 443 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with BPAR in biopsies (following BANFF 2019 criteria) who present Low Sensitivity to the prescribed Immunosupressive drugs in IMBG | 12 months in the prospective follow-up cohort.
  Proportion of patients with BPAR (BANFF 2019 2, 3 or 4) who present Low Sensitivity to the prescribed Immunosupressive drugs in IMBG in longitudinal cohort in 1 year- Protocol Biopsies or in Indication Biopsies and in the cross sectional cohort in Indication Biopsies

SECONDARY OUTCOMES:
Proportion of patients with impairment in renal function AND BPAR or inflammatory damage in biopsies or the presence of dnDSA in the last determination who present low sensitivity to the individual immunosuppressive drugs in IMBG | 12 months
  Proportion of patients with impairment in renal function AND signs of rejection (BPAR) or inflammatory damage in protocol/indication biopsies or the presence of de novo antidonor specific antibodies (dnDSA) in the last determination prior to the biopsy who present low sensitivity to individual prescribed immunosuppressive drugs in IMBG
Proportion of patients with impairment in renal function AND BPAR or inflammatory damage in biopsies or the presence of dnDSA in the last determination who present low sensitivity to all prescribed immunosuppressive drugs in IMBG | 12 months
  Proportion of patients with impairment in renal function AND signs of rejection (BPAR) or inflammatory damage in protocol/indication biopsies or the presence of de novo antidonor specific antibodies (dnDSA) in the last determination prior to the biopsy who present low sensitivity to all prescribed immunosuppressive drugs in IMBG
Proportion of patients with therapeutical failure due to rejection who present low sensitivity to the prescribed immunosuppressive drugs in IMBG | 12 months in the prospective follow-up cohort.
  Proportion of patients with therapeutical failure due to rejection who present low sensitivity to the prescribed immunosuppressive drugs in IMBG (Therapeutical failure is defined as the incidence of graft loss and/or BPAR and/or dnDSA)
Proportion of patients with with therapeutical failure due adverse effects attributable to immunosuppression who present high sensitivity /or low sensitivity and high doses to the prescribed immunosuppressive drugs in IMBG | 12 months in the prospective follow-up cohort.
  Proportion of patients with therapeutical failure due adverse effects attributable to immunosuppression who present high sensitivity /or low sensitivity and high doses to the prescribed immunosuppressive drugs in IMBG Therapeutical failure is defined as the incidence of opportunistic infection by Cytomegalovirus (CMV) (symptomatic or not) and/or BK polyomavirus (BKV) and/or 3 or more hospitalizations due to infections during the patient's follow-up).
Proportion of patients whose pre-transplant IMBG predicts the incidence of events during the patients' follow up | 12 months
  Proportion of patients whose pre-transplant IMBG predicts the incidence of events (graft rejection failure or failure due to adverse effects attributable to immunosuppression) during the patients' follow up
Correlation between IMBG values and other lymphocyte activation markers | In the prospective cohort at 3, 6, 9, and 12 months
  Correlation between IMBG values and other lymphocyte activation markers (CD69, CD25) for each immunosuppressive drug tested with IMBG over time
Distribution of pre-transplant IMBG values and post-transplant at 3, 6, 9, and 12 months | In the prospective cohort at 3, 6 , 9 and 12 months
  Distribution of pre-transplant IMBG values and post-transplant at 3, 6, 9, and 12 months
Adherence to treatment measured with Morisky Green Scale (MMAS). | at 6 and at 12 months
  Adherence to treatment measured with Morisky Green Scale (MMAS, score 0 (worst adherence) - 4 (best adherence), at 6 months and at one year.
Quality of Life perceived by the patient, measured with EQ-5D-5L questionnaire. | baseline and at 12 months
  Quality of Life perceived by the patient, measured with European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) questionnaire (score 0 (worst health) - 100 (best health) at baseline and at one year.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Portero, Study Chair — Biohope Scientific Solutions for Human Health, S.L.
Locations (15):
- Hospital Do Rim, Brasil, Brazil
- University Hospital Grenoble, Grenoble, France
- Germany (2):
  - Charité Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Heidelberg, Heidelberg
- Spain (10):
  - Fundació Puigvert, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Dr. Peset, Valencia
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Portoles JM, Jimenez C, Janeiro D, Lopez-Oliva MO, Ortega-Carrion A, Blanquez D, Arribas L, Gomez C, Diez T, Pascual J, Portero I. The Immunobiogram, a Novel In Vitro Assay to Evaluate Treatment Resistance in Patients Receiving Immunosuppressive Therapy. Front Immunol. 2021 Jan 25;11:618202. doi: 10.3389/fimmu.2020.618202. eCollection 2020. PMID 33569062
- [Background] Pascual J, Jimenez C, Krajewska M, Seron D, Kotton CN, Portoles J, Witzke O, Sorensen SS, Andres A, Crespo M, Paz-Artal E, Diez T, Ortega A, Portero I. The Immunobiogram, a novel in vitro diagnostic test to measure the pharmacodynamic response to immunosuppressive therapy in kidney transplant patients. Transpl Immunol. 2022 Dec;75:101711. doi: 10.1016/j.trim.2022.101711. Epub 2022 Sep 9. PMID 36096417
- [Background] Pascual J, Crespo M, Portoles J, Jimenez C, Ortega-Carrion A, Diez T, Portero I. The IMBG Test for Evaluating the Pharmacodynamic Response to Immunosuppressive Therapy in Kidney Transplant Patients: Current Evidence and Future Applications. Int J Mol Sci. 2023 Mar 8;24(6):5201. doi: 10.3390/ijms24065201. PMID 36982276
- See also: Biohope Scientific Solutions for Human Health, S.L. — https://biohope.eu/